CLINICAL TRIAL: NCT02120534
Title: The Predictive Values of Serum Soluble CD14 Subtype and CD88 Monitoring in Critically Ill Patients.
Brief Title: Serum CD14 and CD88 Mointoring in ICU
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant professor, Tanta University
Other Study IDs: 1638/02/13
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Sepsis
Keywords: soluble CD14 ,serum CD88,sepsis , SIRS.
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis group: Forty seven patients are critically ill with evidence of sepsis during ICU stay (sepsis group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of CD 14 and CD88 will be monitored.
- SIRS group: Forty seven patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of CD 14 and CD88 will be monitored.

SUMMARY:
The present study will be conducted to determine the dynamic changes of serum soluble CD14 and the corresponding changes of serum CD88 and their correlation in critically ill sepsis and SIRS patients.

DETAILED DESCRIPTION:
A total of ninty four will be included in the study. Forty seven patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and forty seven patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of CD 14 and CD88 will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* The patients staying in ICU for more than 24 hours will be included in the study.

Exclusion Criteria:

* Patients received anti-inflammatory drugs or corticosteroids before admission, patients had immunosuppressive illness, patients had chronic organ failure; patients received massive blood transfusion; patients with radiation therapy and patients with previous organ transplantation will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of ninety-four patients will be included in the study. Forty seven patients are critically ill with evidence of sepsis during ICU stay (sepsis group) and forty seven patients are critically ill without evidence of infectious organism (SIRS group). At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of CD 14 and CD88 will be monitored.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
A serum soluble CD14 | one week
  At admission, Patients data include clinical status; SOFA score; central venous pressure; laboratory analysis and arterial blood gas analysis are measured. Routine cultures will be obtained. The attending physician will evaluate the patients for sepsis, severe sepsis, or septic shock as long as their stay in ICU. A serum level of CD 14 will be monitored.

SECONDARY OUTCOMES:
Survival of ICU patients | Two weeks
  Correlation of of serum soluble CD14 and the corresponding changes of serum CD88 and their correlation in critically ill sepsis and SIRS patients and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant Professor
Locations (1):
- Tanta University Hospitals, Tanta, Algharbyia, Egypt